CLINICAL TRIAL: NCT00004883
Title: A Phase II Trial of Trastuzumab (Herceptin) for Advanced Stage (IIIB, IV), HER2 Overexpressing, Non-Small Cell Lung Cancer
Brief Title: Trastuzumab in Treating Patients With Stage IIIB or Stage IV Non-small Cell Lung Cancer That Overexpresses HER2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02318; CLB-39810; U10CA031946 (NIH); CDR0000067555 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-03-07; First posted 2003-09-30 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Recurrent Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Trastuzumab

ARMS (1):
- Treatment (trastuzumab) (Experimental): Patients receive trastuzumab (Herceptin) IV over 30-90 minutes on day 1. Treatment continues once a week in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: trastuzumab; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: trastuzumab — Given IV
  Other Names: anti-c-erB-2; Herceptin; MOAB HER2
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of trastuzumab in treating patients who have stage IIIB or stage IV non-small cell lung cancer that overexpresses HER2. Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the activity of trastuzumab (Herceptin) in patients with stage IIIB or IV HER2-overexpressing non-small cell lung cancer.

SECONDARY OBJECTIVES:

I. Determine the duration of response in patients treated with this regimen. II. Determine the toxicity of this treatment regimen in this patient population.

III. Assess levels of circulating HER2 and correlate with HER2 expression in this patient population.

V. Correlate circulating HER2 levels with non-small cell lung cancer tissue HER2 expression.

OUTLINE:

Patients receive trastuzumab (Herceptin) IV over 30-90 minutes on day 1. Treatment continues once a week in the absence of disease progression or unacceptable toxicity.

Patients are followed every 8 weeks until disease progression or death.

PROJECTED ACCRUAL: Approximately 84 patients (42 per stratum) will be accrued for this study within 17.5 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage IIIB or IV non-small cell lung cancer

  * Supraclavicular node involvement allowed
  * Malignant pleural effusion allowed (cytological confirmation not required if pleural fluid bloody or exudative)
* No stage IIIB patients eligible for CLB protocols comprising combined chemotherapy and chest radiotherapy
* Recurrent disease allowed
* HER2 overexpression (2-3+)
* At least 1 unidimensionally measurable lesion

  * At least 20 mm by conventional techniques
  * At least 10 mm by spiral CT scan
  * The following are not considered measurable:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Abdominal masses not confirmed and followed by imaging
    * Cystic lesions
* No CNS metastases
* Performance status - ECOG 0-2
* Granulocyte count at least 1,500/mm3
* Platelet count at least 100,000/mm3
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* Creatinine no greater than 1.5 times ULN
* LVEF at least 45% (by echocardiogram or MUGA)
* Not pregnant or nursing
* Fertile patients must use effective contraception
* HIV negative
* No concurrent immunologic disease (e.g., autoimmune disease)
* No history of allergy to murine products
* No prior murine antibodies
* No prior anthracyclines
* No more than 1 prior chemotherapy regimen for lung cancer
* At least 4 weeks since prior chemotherapy
* No concurrent chemotherapy
* No concurrent steroids except for adrenal failure or dexamethasone as an antiemetic
* No concurrent hormonal therapy except for nondisease-related conditions (e.g., insulin for diabetes)
* At least 6 months since prior radiotherapy
* No concurrent palliative radiotherapy
* At least 4 weeks since prior major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2000-02; Primary Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Response rate (complete response [CR] and partial response [PR]) | Up to 5 years

SECONDARY OUTCOMES:
Overall survival (OS) | From registration until death or last known follow-up, assessed up to 5 years
  Kaplan-Meier curves will be used to describe OS.
Failure-free survival (FFS) | Time between registration and disease progression, death, or last known follow-up, assessed up to 5 years
  Kaplan-Meier curves will be used to describe FFS.
Duration of response | Time between the initial documentation of response and subsequent failure (death, disease progression), assessed up to 5 years
  Kaplan-Meier curves will be used to describe duration of response.
Toxicity as assessed by NCI's Common Toxicity Criteria | Up to 5 years
  The frequency of occurrence of various toxicities will be tabulated by the most severe occurrence experienced by each individual patient.
Relationship between HER2 expression in tumor tissue and serum | Up to 5 years
  A 95% confidence interval for this proportion will be estimated using the binomial distribution. The level of circulating HER2 receptor will be descriptively summarized with means, medians, quartiles, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Clamon, Principal Investigator — Cancer and Leukemia Group B
Locations (1):
- Cancer and Leukemia Group B, Chicago, Illinois, United States